CLINICAL TRIAL: NCT04395820
Title: Prospective Surveillance of Lung Development During Childhood, Adolescence and Adulthood in Healthy and Patients With Cystic Fibrosis
Acronym: Prospective
Status: Active, not recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Kathryn Ramsey, Principal Investigator, Insel Gruppe AG, University Hospital Bern
Other Study IDs: 2019-01591
Record Dates: First submitted 2020-05-05; First posted 2020-05-20 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Cystic Fibrosis; Healthy
Keywords: Cystic Fibrosis; MBW; MRI; Airway growth; Airway development; Healthy
MeSH Terms: conditions — Cystic Fibrosis | interventions — Respiratory Function Tests; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oropharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis
  Interventions: Diagnostic Test: Lung function test; Diagnostic Test: Imaging
- Healthy
  Interventions: Diagnostic Test: Lung function test; Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Lung function test — MBW
Diagnostic Test: Imaging — MP-MRI

SUMMARY:
Cystic fibrosis (CF) is the most common lethal inherited disease in Caucasian populations. To improve survival, it is essential to understand the development, progression and treatment of CF lung disease throughout early childhood.

Therefore the overall objective is to prospectively assess the clinical utility of novel and non-invasive measuring methods, namely Multiple Breath Washout and functional lung MRI in the longitudinal clinical surveillance of patients with CF and compare the results to those of healthy controls.

DETAILED DESCRIPTION:
Background and project rationale:

Cystic fibrosis (CF), the most common lethal inherited disease in Caucasian populations, affects approximately 1:2500 live births. It is a multisystem disorder with respiratory morbidity and mortality being the leading cause of death. Despite improved survival in successive birth cohorts, the current median survival age of patients with CF is about 40 years. To improve survival, it is essential to understand the development, progression and treatment of CF lung disease throughout early childhood. Therefore tracking of lung function throughout childhood may provide important insights into the development and progression of CF lung disease. Spirometry, the standard lung function test for decades, is sensitive only for airflow limitation arising in large airways and insensitive for assessment of small or peripheral airway involvement, whereby the CF lung disease emerges in the small airways. Two promising techniques to assess small airway function in young children include the multiple breath washout (MBW) lung function test and functional Matrix-Pencil magnetic resonance imaging (MP-MRI).

Project Objectives and Design:

The overall objective of this project is to prospectively assess the clinical utility of MBW and MP-MRI in the longitudinal clinical surveillance of patients with CF. Therefore this study: i) Examines differences in MBW and MP-MRI outcomes between patients with CF and healthy controls. ii) Assesses the short term (over 1h) repeatability of MBW and MP-MRI outcomes in patients with CF and healthy controls. iii) Assesses whether MBW and MP-MRI outcomes are associated with clinical lung disease in patients with CF. iv) Determines whether changes in MBW and MP-MRI outcomes are associated with progression of lung disease in patients with CF. v) Compares the breath-by-breath regional and temporal changes in functional MRI signal with breath-by-breath changes in MBW phase outcomes in patients with CF and healthy controls.

Methods:

Data of MBW, MP-MRI, morphological MRI, Spirometry and body plethysmography, clinical respiratory symptoms and microbiology will be collected during this study.

Recruitment and participation:

Children and adults with CF will be recruited from the outpatient and inpatient clinics at the Inselspital in Bern. Healthy controls will be recruited from the local community in Bern and surrounding areas.

Information collected:

Lung function:

* Multiple Breath Washout (FRC, LCI, Scond, Sacin)
* Spirometry (FEV1, FVC, FEFx)
* Body plethysmography (sReff, FRCpletz, TLC)

Respiratory symptoms and clinical data:

CF:

* respiratory symptoms (cough, sputum characteristics, shortness of breath, weight loss, appetite fatigue)
* clinical data (increased work of breathing, hypoxemia, wheeze, crackles, differential air entry)

Healthy controls:

Presence of respiratory symptoms in the last four weeks preceding visit.

Functional and structural MRI:

* Functional MRI (percentage of the lung volume with impaired fractional ventilation (RFV) and relative perfusion (RQ)
* Structural MRI( Eichinger MRI scoring system to assess the presence and extent of bronchiectasis, mucous plugging, and air trapping)

Medical history:

CF: demographics, genetic mutation, pulmonary exacerbations, hospitalisations, regular therapy and medication, complications, microbiological data and laboratory reports

Microbiology:

CF: bacterial analysis of oropharyngeal swabs

Quality of life:

CF: CF-specific quality of life and symptoms

Sputum:

CF:

* spontaneously expectorated sputum
* Induced sputum

Study database:

All study data is recorded in an Access-database with SQL Servers. The database is accordant to the HFG and was adapted together with the CTU.

Funding:

The Swiss National Foundation (32003B_182719) and Vertex-Pharmaceuticals Cystic Fibrosis Research Innovation Award provide financial and material support for this observational study

ELIGIBILITY:
Inclusion Criteria:

Individuals with CF:

* Diagnosis of CF
* Signed written informed consent
* ≥3 - 18 years of age, depending on the cooperation and if lung function measurements are possible

Healthy volunteers:

* Signed written informed consent
* Informed consent of participant and if under 18 years, legal representative respectively
* Children and adults with no history of chronic lung disease or acute respiratory infection in the four weeks prior to the study visit
* ≥3 - 18 years of age, depending on the cooperation and if lung function measurements are possible

Exclusion Criteria:

The presence of any one of the following exclusion criteria will lead to exclusion of the participant, for example:

* Women who are pregnant or breast feeding.
* Intention to become pregnant during the course of the study
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Please note that female participants who are surgically sterilised/hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Other clinically significant concomitant disease states (e.g. renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Known or suspected non-compliance, drug or alcohol abuse
* Continuous glucose monitor
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, etc. of the participant
* Metal in body, e.g. pacemaker
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Subjects which are respiratory insufficient to attend on the lung function measurements (oxygen demand)
* Subjects who are unable to perform the MRI without sedation
* Participants which were born preterm (<36. week of pregnancy)
* Current smokers

In addition for individuals with CF:

* Known diseases other than related to CF

In addition for healthy individuals:

* Current upper respiratory infection (cough, cold, fever) will lead to postponement of the visit to 4 weeks after the end of symptoms

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adults with CF and healthy volunteers from the local community in Bern and surrounding areas.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2050-12-01 (Estimated); Study Completion 2100-12-01 (Estimated)

PRIMARY OUTCOMES:
Multiple Breath Washout | Every third month up to 50 years. Healthy controls only during 1 year.
  Longitudinal assessment of lung volume and ventilation inhomogeneity
Functional MP-MRI | Every twelfth month up to 50 years. Healthy controls only during 1 year (2 time points).
  Longitudinal assessment of percentage of the lung volume with impaired fractional ventilation and relative perfusion

SECONDARY OUTCOMES:
Morphological MRI | Every twelfth month up to 50 years. Healthy controls only during 1 year (2 time points)
  Longitudinal assessment of the presence and extent of bronchiectasis, mucous plugging and air trapping by Eichinger MRI scoring.
Spirometry: FEV1 | Every third month up to 50 years. Healthy controls only during 1 year.
  Longitudinal assessment of forced expired volume in 1 second.
Spirometry: FVC | Every third month up to 50 years. Healthy controls only during 1 year.
  Longitudinal assessment of forced vital capacity.
Spirometry: FEF | Every third month up to 50 years. Healthy controls only during 1 year.
  Longitudinal assessment of forced expiratory flows.
Body plethysmography: sRAW | Every third month up to 50 years. Healthy controls only during 1 year.
  Longitudinal assessment of specific airway resistance.
Body plethysmography: FRC | Every third month up to 50 years. Healthy controls only during 1 year.
  Longitudinal assessment of functional residual capacity.
Body plethysmography: TLC | Every third month up to 50 years. Healthy controls only during 1 year.
  Longitudinal assessment of total lung capacity.
Respiratory symptoms | Every third month up to 50 years. Only CF patients.
  Longitudinal assessment of clinical respiratory symptoms.
Exacerbations | Every third month up to 50 years. Only CF patients.
  Longitudinal assessment of clinical status.
CF-related quality of life | Every third month up to 50 years. Only CF patients.
  Longitudinal assessment of standardised age-specific CF-related quality of life questions.The scale goes from 0-100, higher score means better outcome.
Microbiology: presence of respiratory pathogens | Every third month up to 50 years. Only CF patients.
  Longitudinal assessment of presence of respiratory pathogens from oropharyngeal swabs and sputum samples.
Microbiology: abundance of respiratory pathogens | Every third month up to 50 years. Only CF patients.
  Longitudinal assessment of abundance of respiratory pathogens from oropharyngeal swabs and sputum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Ramsey, PhD, Principal Investigator — University Children's Hospital Bern
Locations (1):
- University Children's Hospital Bern, Bern, Switzerland

REFERENCES:
- [Background] O'Sullivan BP, Freedman SD. Cystic fibrosis. Lancet. 2009 May 30;373(9678):1891-904. doi: 10.1016/S0140-6736(09)60327-5. Epub 2009 May 4. PMID 19403164
- [Background] Ramsey KA, Ranganathan S, Park J, Skoric B, Adams AM, Simpson SJ, Robins-Browne RM, Franklin PJ, de Klerk NH, Sly PD, Stick SM, Hall GL; AREST CF. Early respiratory infection is associated with reduced spirometry in children with cystic fibrosis. Am J Respir Crit Care Med. 2014 Nov 15;190(10):1111-6. doi: 10.1164/rccm.201407-1277OC. PMID 25321321